CLINICAL TRIAL: NCT06572878
Title: Evaluation of the Effect of Cognitive and Physical Training on Mild Cognitive Impairment Elder's Physical and Cognition Domain: A Clinical Trial.
Brief Title: Evaluation of Cognitive and Physical Training on MCI Elders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Jia-You, YE, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202404122
Record Dates: First submitted 2024-08-01; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Impairment; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive training (Experimental): Each participant will receive cognitive training for 45 minutes per session, three sessions per week, for 12 weeks.
  Interventions: Other: Cognitive training
- Physical training (Experimental): Each participant will receive physical training for 45 minutes per session, three sessions per week, for 12 weeks.
  Interventions: Other: Physical training
- Combined cognitive and physical training (Experimental): Each participant will receive combined cognitive and physical training for 45 minutes per session, three sessions per week, for 12 weeks.
  Interventions: Other: Combined cognitive and physical training
- Passive information activities (Active Comparator): Each participant will engage in passive information activities for 45 minutes per session, three sessions per week, for 12 weeks.
  Interventions: Other: Passive information activities

INTERVENTIONS:
Other: Cognitive training — Cognitive training will follow a group format, with each group consisting of 4-16 participants. Each group will be in a private, independent room for their training sessions and will not interact with participants from other groups. The cognitive training task components will specifically focus on attention, learning and memory, executive function, perceptual-motor skills, and language.
  Arms: Cognitive training
Other: Physical training — Physical training will follow a group format, with each group consisting of 4-16 participants. Each group will be in a private, independent room for their training sessions and will not interact with participants from other groups. The physical training task components will specifically focus on strength, balance, agility, gait, low-volume aerobic, and flexibility.
  Arms: Physical training
Other: Combined cognitive and physical training — Combined cognitive and physical training will follow a group format, with each group consisting of 4-16 participants. Each group will be in a private, independent room for their training sessions and will not interact with participants from other groups. The combined cognitive and physical training components will specifically focus on a single cognitive task and simultaneously handle a single physical task.
  Arms: Combined cognitive and physical training
Other: Passive information activities — In passive informational activities, which include a variety of puzzles, audiobooks, and diverse reading materials such as newspapers or listening to news content.
  Arms: Passive information activities

SUMMARY:
This study examines the impact of combining cognitive and physical training, recognizing that daily living often requires individuals to perform multiple tasks simultaneously. The inability to execute such dual movements can hinder daily functioning.

The primary goal is to enhance the ability of individuals with mild cognitive impairment (MCI) to perform two tasks concurrently, focusing on both cognitive and physical aspects. This research aims to deepen our understanding of how multitasking affects patients' abilities and to develop effective intervention programs.

DETAILED DESCRIPTION:
The World Health Organization has recognized cognitive impairment as a significant global health issue, encompassing a spectrum of conditions from mild cognitive impairment to various forms of dementia. These conditions are linked to heightened risks of disability and mortality. In the absence of suitable interventions, cognitive functions typically exhibit a gradual decline over time, driven by factors including aging, neurological disorders, traumatic brain injury, and substance abuse.

A thorough literature review indicates that cognitive and physical training can sustain cognitive or physical functions, contingent upon the specific training protocols implemented. Concurrent cognitive and physical training entails the simultaneous execution of multiple cognitive and motor activities, thereby maintaining dual functional control. This innovative training modality integrates motor and cognitive rehabilitation into a cohesive framework.

This clinical trial adopts a randomized controlled design, stratifying participants into four distinct groups: cognitive training, physical training, combined cognitive and physical training, and passive informational activities. The interventions will be administered with a frequency of three times per week over a 12-week period, incorporating task-specific training to enhance both motor and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged 60 years or older and able to communicate in Mandarin or Taiwanese.
2. Mild cognitive impairment, assessed using the Mini Mental State Examination (MMSE) with a score of 14≦MMSE≦25.
3. Self-reported complaints of cognitive decline.
4. In addition to the above criteria, participants must voluntarily agree to participate and sign an informed consent form.

Exclusion Criteria:

1. Individuals with severe psychiatric disorders or behavioral problems, as assessed by the Neuropsychiatric Inventory Questionnaire (NPI-Q) with (a) severity score ≥ 6 and caregiver distress score ≥ 7.
2. Participants who have undergone other cognitive or activity training within the past six months.
3. Individuals with sensory impairments, such as visual, auditory, or communication difficulties.
4. People with mobility impairments, such as those who use wheelchairs or mobility aids.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  The Mini-Mental State Examination (MMSE) is a standardized instrument for assessing overall cognitive function, where higher scores indicate better global cognition, with a total score ranging from 0 to 30. It is crucial to consider both age and education levels when interpreting the results.
Wisconsin Card Sorting Test - Computer Version | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  The Wisconsin Card Sorting Test (WCST) is a standardized instrument for assessing executive function. Interpreting WCST results includes analyzing the total correct responses and total errors. The total correct responses indicate the number of correct matches made by the participant; a higher number of correct responses suggests better overall cognitive performance and the ability to learn and apply the rules. Conversely, a high number of errors can indicate difficulties in understanding or applying the sorting rules.
Digit Span Test | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  A standardized instrument for assessing working memory.
Shor-form Berg balance scale | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  The Short-Form Berg Balance Scale (SFBBS) is a streamlined assessment tool designed to evaluate an individual's balance and stability. Each item on the SFBBS is scored on a scale from 0 to 4, with 0 indicating the lowest level of function and 4 indicating the highest level of function. The scores for each item are summed to obtain a total score, which provides an overall measure of balance. The maximum possible score varies depending on the number of items included in the short form.
Back scratch test | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  A flexibility test.
Chair sit-and-reach test | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  A flexibility test.
Grip and pinch strength | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  A standardized instrument " PABLO®" for assessing strength.
Gait analysis | Baseline, 6 weeks (mid), 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  A standardized instrument " PABLO®" for assessing gait performance.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized instrument for assessing sleep quality and disturbances over a 1-month period. It evaluates seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction during the month preceding the test. The total score ranges from 0 to 21 points, with a total score greater than 5 indicating poor sleep.
Insomnia Severity Index | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  The Insomnia Severity Index (ISI) is a validated tool for assessing the severity of insomnia symptoms and their impact on daily functioning. The scores for each item are summed to obtain a total score, which ranges from 0 to 28, with higher scores indicating worse sleep. A total score greater than 8 suggests the presence of insomnia.
Actigraphy sleep efficiency (%) | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  Sleep parameters were measured using wrist actigraphy (GT9X; Manufacturing Technology, Pensacola, FL, USA) to collect sleep data. Mean sleep efficiency was derived from actigraphy recordings as the ratio of total sleep time to time in bed, multiplied by 100. Restlessness, indicated by a sleep efficiency below 80%, should be carefully considered in elderly individuals.
Actigraphy total sleep time (minutes) | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  Sleep parameters are measured by the wrist actigraphy (GT9X; Manufacturing Technology, Pensacola, FL, USA) to collect sleep data. Mean total sleep time derived from actigraphy recordings.
Actigraphy wake duration (minutes) | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  Sleep parameters are measured by the wrist actigraphy (GT9X; Manufacturing Technology, Pensacola, FL, USA) to collect sleep data. Mean wake after sleep onset derived from actigraphy recordings.
Actigraphy sleep onset latency (minutes) | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  Sleep parameters are measured by the wrist actigraphy (GT9X; Manufacturing Technology, Pensacola, FL, USA) to collect sleep data. Mean sleep onset latency derived from actigraphy recordings. Restlessness, indicated if more than 30-60 minutes, should be carefully considered in elderly individuals.
Actigraphy time in bed (minutes) | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  Sleep parameters are measured by the wrist actigraphy (GT9X; Manufacturing Technology, Pensacola, FL, USA) to collect sleep data. Mean time in bed derived from actigraphy recordings.
Actigraphy sleep fragmentation (%) | Baseline, 12 weeks (post-intervention), 3 months, and 6 months after completing the intervention
  Sleep parameters are measured by the wrist actigraphy (GT9X; Manufacturing Technology, Pensacola, FL, USA) to collect sleep data. Sleep fragmentation index (sum of limb movement and fragmentation indexes). The restlessness index during sleep, expressed as a percentage, indicates sleep disruption; higher values mean more disrupted sleep.

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data (IPD) available to other researchers.